CLINICAL TRIAL: NCT00132847
Title: German Cockroach Allergen Standardization Evaluation (CASE)
Brief Title: Comparing Allergenic Effects of 3 German Cockroach Extracts in Adults
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-03
Record Dates: First submitted 2005-08-08; First posted 2005-08-22 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Asthma; Allergy
Keywords: Child; Adolescent; Urban Health
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: German Cockroach Allergen extract

SUMMARY:
The purpose of this study is to test and compare the allergenic effects of three commercially available German cockroach allergen extracts in adults.

Study hypothesis: The biological potency of three commercially available German cockroach allergy extracts can be compared using the ID50EAL method to standardize German cockroach allergens.

DETAILED DESCRIPTION:
Cockroach allergens appear to be a major cause of inner city asthma. Because of the suspected relationship between domestic cockroach species and allergy and asthma symptoms, the Food and Drug Administration (FDA) wants to standardize cockroach allergen vaccines for use in the U.S. Allergen standardization comprises two important components: the selection of a reference preparation of allergenic extract and the selection of procedures to compare manufactured products to the reference allergen extract.

Adults in this study will be exposed to different doses of each of 3 German cockroach allergen extracts via intradermal skin testing. Participants in this study will be adults who have a history of allergic disease or asthma and are sensitive to the German cockroach allergens being tested.

Participants will have 2 visits during this study: a screening session and a testing session. At screening, participants will be asked to complete a screening questionnaire and will undergo a targeted physical exam, vital signs measurement, and peak expiratory flow (PEF) testing. Premenopausal women will also have urine collected for pregnancy testing. At the screening session, a 15-minute prick/puncture test will be administered on the skin of the forearm with the proposed standard allergen extract, histamine (positive control), and diluent (negative control). Skin erythema (swelling) response to the injections will be recorded.

Some participants may continue into the testing session on the same day as the screening session; others will participate in the testing session at a second study visit within 4 weeks after study screening. At the start of the testing session, participants will be asked to complete a questionnaire about demographics, history of airway disease and previous skin testing, and current medication use. For participants whose testing session occurs on a different day than the screening session, vital signs measurement and PEF readings will occur and premenopausal women will have urine collected. Blood collection will occur prior to the skin test. Intradermal skin testing will consist of injections on the participant's back with multiple doses of 3 different extracts of German cockroach allergen. Each of the 3 extracts will require 4 to 7 injections, depending on the response to each dose. Erythema skin response to the dilutions will be recorded. Participants will be observed for at least 1 hour after the intradermal skin testing as a safety precaution. After the observation period, participants will undergo additional PEF testing and will be assessed for adverse reactions to the skin testing procedure. Participants may be given antihistamines to relieve itching.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Speak English
* Have valid prick/puncture skin test defined by sum of erythema to histamine base (1.0 mg/ml) of 35 mm or greater
* Have intradermal skin test defined by sum of erythema to histamine base (0.275 mg/ml : 0.1 mg/ml base) of 35 mm or greater
* Self-reported history of allergic disease, such as symptoms compatible with allergic rhinitis or asthma
* Erythema diameter response of 30 mm or greater to a prick/puncture skin test with an undiluted preparation of one of the cockroach allergen extracts being tested
* Available for the duration of the study

Exclusion Criteria:

* Skin coloring or condition that would complicate the measurement of erythema responses
* Dermographism (development of hives following skin contact with an object) greater than a 4 mm erythema diameter response following saline skin test at screening
* Current use of tricyclic antidepressants, MAO inhibitors, or beta-blockers
* Current use of antihistamines
* Use of topical steroids in the 14 days prior to study screening on the areas to be skin tested
* Current use of oral or parenteral corticosteroids
* Current use of inhaled steroids. More information on this criterion can be found in the protocol.
* Unable to provide a contact name in case of an emergency
* History of anaphylaxis
* Have been to the emergency room for asthma within the last month prior to study entry
* Hospitalization for asthma within the last 6 months prior to study entry
* Cardiovascular disease. Participants who have had mitral valve prolapse or who have well-controlled hypertension are not excluded.
* Pregnant or breastfeeding
* Peak expiratory flow (PEF) of less than 75% predicted at screening or testing sessions
* Past or present immunotherapy with the test allergen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a group of adults who have a history of allergic disease or asthma and demonstrate sensitivity to the German cockroach allergen being tested
Enrollment: 4 (Actual)
Dates: Start 2004-04; Study Completion 2004-10

PRIMARY OUTCOMES:
Biological potency of three commercially available German cockroach allergen extracts
  measured in units of BAU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Peyton Eggleston, MD, Principal Investigator — Johns Hopkins University; Jacqueline Pongracic, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Stan Szefler, MD, Principal Investigator — National Jewish Health; Floyd Malveaux, MD, PhD, Principal Investigator — Howard University; William W. Busse, MD, Study Director — University of Wisconsin, Madison

REFERENCES:
- [Background] Arruda LK, Ferriani VP, Vailes LD, Pomes A, Chapman MD. Cockroach allergens: environmental distribution and relationship to disease. Curr Allergy Asthma Rep. 2001 Sep;1(5):466-73. doi: 10.1007/s11882-001-0035-1. PMID 11892074
- [Background] Arruda LK, Vailes LD, Ferriani VP, Santos AB, Pomes A, Chapman MD. Cockroach allergens and asthma. J Allergy Clin Immunol. 2001 Mar;107(3):419-28. doi: 10.1067/mai.2001.112854. PMID 11240940
- [Background] Eggleston PA. Environmental causes of asthma in inner city children. The National Cooperative Inner City Asthma Study. Clin Rev Allergy Immunol. 2000 Jun;18(3):311-24. doi: 10.1385/CRIAI:18:3:311. No abstract available. PMID 10981263
- [Background] Patterson ML, Slater JE. Characterization and comparison of commercially available German and American cockroach allergen extracts. Clin Exp Allergy. 2002 May;32(5):721-7. doi: 10.1046/j.1365-2222.2002.01397.x. PMID 11994096